CLINICAL TRIAL: NCT06191952
Title: Davos Alzheimer's Collaborative Healthcare System Preparedness to Increase Cognitive Assessment Rates for Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: ki:elements (Unknown); Hoffmann-La Roche (Industry); Eisai Limited (Industry); Johanniter-Unfall-Hilfe e.V. (Unknown); University of Southern California (Other)
Responsible Party: Principal Investigator, Robert Perneczky, Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 22-0786
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Subjective Cognitive Decline; Alzheimer Dementia
Keywords: Subjective Cognitive Decline; Mild Cognitive Impairment; Community Setting; Digital Cognitive Tests; Blood Biomarker
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjective Cognitive Decline Questionnaire (SCD-Q)/no other procedure (Other): Participants will undergo procedure as usual and fill out the questionnaire SCD-Q
  Interventions: Diagnostic Test: Subjective cognitive decline questionnaire (SCD-Q); Diagnostic Test: ki:elements digital speech biomarker for cognition (ki:e SB-C)
- SCD-Q + digital cognitive testing using Cognigram (Other): Participants will undergo procedure as usual with their GP, additionally they will fill out the SCD-Q and undergo cognitive testing (Cognigram)
  Interventions: Diagnostic Test: Cognigram; Diagnostic Test: Subjective cognitive decline questionnaire (SCD-Q); Diagnostic Test: ki:elements digital speech biomarker for cognition (ki:e SB-C)
- SCD-Q + Cognigram + blood-based biomarkers (Other): Participants will undergo procedure as usual with their GP, additionally they will fill out the SCD-Q and undergo cognitive testing (Cognigram). The blood-based biomarkers will be determined.
  Interventions: Diagnostic Test: Cognigram; Diagnostic Test: Subjective cognitive decline questionnaire (SCD-Q); Diagnostic Test: blood-based biomarkers; Diagnostic Test: ki:elements digital speech biomarker for cognition (ki:e SB-C)

INTERVENTIONS:
Diagnostic Test: Cognigram — Cognigram (previously known as the Cogstate Brief Battery) is a brief, computer-administered cognitive test battery requiring about 20-25 minutes for administration, consisting of four cognitive tasks to measure psychomotor function, attention, working memory, and learning and memory. Eisai owns the commercial rights for Cognigram and has kindly agreed to offer the required licenses for the present project free of charge. Digital cognitive testing will take place in the respective social and care centers on a tablet which is not connected to the internet. Testing will be performed pseudonymized and data from the cognitive tests will be downloaded regularly by the study team and added to the database at LMU hospital.
  Arms: SCD-Q + Cognigram + blood-based biomarkers; SCD-Q + digital cognitive testing using Cognigram
Diagnostic Test: Subjective cognitive decline questionnaire (SCD-Q) — The SCD-Q is a validated questionnaire assessing the presence of subjective cognitive deterioration in abilities such as memory, attention, language, and executive function. The scale includes 24 dichotomous questions (yes/no), evaluating decline in daily life during the last two years. The SCD-Q score ranges from 0 to 24, with higher scores indicating greater perceived cognitive change (cut-off classified as SCD equal or greater as 7).
Diagnostic Test: blood-based biomarkers — Blood plasma and serum samples will be collected by the project staff according to standard operating procedures used at LMU Munich and subsequently processed and measured at the Department of Psychiatry and Psychotherapy to quantify the blood-based biomarkers for AD using Elecsys immunoassays running on a Cobas e402 analyzer. All test results (including the respective cut-off measurements for normal vs abnormal) will be forwarded directly to the participants' GPs. No further explanations and instructions will be provided to avoid any unwanted bias, and participants will only be informed about their results by their doctors. Roche has kindly offered to provide blood biomarker assays free of charge for the present project.
  Arms: SCD-Q + Cognigram + blood-based biomarkers
Diagnostic Test: ki:elements digital speech biomarker for cognition (ki:e SB-C) — The ki:elements digital speech biomarker for cognition (ki:e SB-C) can be collected remotely in fully automated telephone visits, taking 15 minutes to complete based on three specific assessments measuring learning and memory, processing speed, executive function, and language capabilities. The ki:e SB-C uses artificial intelligence and automatic speech analysis to process and transcribe speech, followed by an extraction of relevant features, combined into four subdomain and one global cognition score.

SUMMARY:
In this study the investigators explore a pragmatic strategy to increase cognitive screening rates in the community. The investigators will compare the monetary value of different combinations of SCD questionnaires, digital cognitive tests, and blood Alzheimer's Disease (AD) biomarkers to identify the best approach for primary care settings.

DETAILED DESCRIPTION:
The investigators aim to perform a cluster-randomized study, exploring the effectiveness, efficiency, and acceptability of a pragmatic strategy to increase cognitive screening rates in the community. Participants will be older adults attending social and cultural centers in the greater Munich area. The investigators will compare the monetary value of different combinations of SCD questionnaires, digital cognitive tests, and blood AD biomarkers to identify the best approach for primary care settings. As secondary aims, qualitative interviews will be conducted with general practitioners (GPs) and their patients to explore the acceptability of the proposed new screening strategy; furthermore, the diagnostic utility of an artificial intelligence-based automated analysis of speech will be assessed. The initiative will not only generate novel insights into the optimal approach for large-scale cognitive screening in the general population, but also contribute to an urgently required cultural change in Germany, resulting in a sustainable solution for effective and efficient early recognition and prevention of dementia.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older

Exclusion Criteria:

* younger than 65 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participating individuals screening positive for SCD | Baseline
  The primary endpoint of this protocol is to assess the proportion of participating individuals aged 65 years or older screening positive for SCD during the intervention period who are referred to specialist evaluation, by study arm (intent to treat)

SECONDARY OUTCOMES:
Proportion of individuals with early-stage AD diagnosis | Baseline
  Proportion of individuals formally diagnosed with early-stage AD in a specialist clinic, by study arm
average time to diagnosis of AD | Baseline
  Average time to diagnosis of early-stage AD, by study arm
Qualitative interviews | Baseline
  Qualitative participant and GP interviews on perceived changes/benefits/barriers, lessons learned, etc., per study arm
Correlation with speech analysis and other diagnostic tests | Baseline
  Correlation of ki:e SB-C global and domain cognitive scores with established AD neuropsychological tests and biomarkers (PET, cerebrospinal fluid, blood) and added value of automated speech assessment in routine cognitive assessment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Perneczky, Prof. Dr., Principal Investigator — Klinik und Poliklinik für Psychiatrie und Psychotherapie des LMU Klinikums
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie des LMU Klinikums, München, Bavaria, Germany